CLINICAL TRIAL: NCT00096759
Title: Efficacy of CAM Interventions in Rheumatoid Arthritis
Brief Title: Comparing Tai Chi Chih and Relaxation Therapy in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002307-01 (NIH)
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Tai Chi; Meditation; Relaxation Techniques
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Tai Chi Chih
Behavioral: Relaxation training

SUMMARY:
The purpose of this study is to compare the effectiveness of relaxation therapy and tai chi in treating the symptoms of rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
RA is a debilitating disease characterized by inflammation of the joints, leading to chronic pain, loss of function, and disability. Complementary and alternative medicine (CAM) treatments are being used with increased frequency by patients with chronic pain and rheumatic diseases to relieve their symptoms. While patients find these treatments helpful, there is limited scientific evidence of the effectiveness of these interventions. This study will compare relaxation therapy (a commonly used treatment for RA) to tai chi chih (a combination of slow, deliberate movements and meditation) in treating the symptoms of RA.

Participants will be randomly assigned to receive 12 weeks of either relaxation therapy or tai chi chih. At study entry and Weeks 6 and 12, participants will complete questionnaires about their RA symptoms, health functioning, overall quality of life, and complete a brief medical exam.

ELIGIBILITY:
Inclusion Criteria:

* Active adult onset rheumatoid arthritis
* Stable on disease-modifying antirheumatic drugs (DMARDs) or biologic medications
* Able to walk without use of an assistive device
* Resides in greater Los Angeles area
* Willing and able to comply with study requirements

Exclusion Criteria:

* Uncontrolled or untreated medical conditions
* Frequent or uncontrolled disease flares
* Use of certain medications any medical condition deemed by the investigators to interfere with either the patient's safe participation or interpretation of the study data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
RA-related disability
Health functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Pike, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California